CLINICAL TRIAL: NCT06581146
Title: A Non-interventional, Epidemiologic Study of XLMTM and Clinical Expression in the Liver
Brief Title: A Study to Check Liver Health in Boys With XLMTM, a Serious Genetic Muscle Condition
Acronym: EXCEL
Status: Recruiting | Type: Observational
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 1600-MA-3536
Record Dates: First submitted 2024-08-19; First posted 2024-09-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: X-Linked Myotubular Myopathy
Keywords: XLMTM; Hepatobiliary
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with XLMTM: Pediatric and adolescent participants with XLMTM.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No investigational drug will be administered to participants in this study.

SUMMARY:
XLMTM (X-linked myotubular myopathy) is a serious genetic muscle condition. It is caused by changes in the MTM1 gene which stops or slows down normal muscle development, causing severe muscle weakness. There is currently no cure for XLMTM. Ongoing care is needed to manage symptoms and prevent further medical problems from this condition.

Recent research shows that individuals with XLMTM often have reduced bile flow which can affect liver and gallbladder health. Bile is a liquid made in the liver that helps digest fat. Ongoing liver health checks may help with the routine care of people with XLMTM.

There is a need to understand liver problems that develop in individuals with XLMTM over time. The main aim of the study is to learn how many boys with XLMTM have new cases of liver problems during the study.

This study is about collecting information only. This is known as an observational study. The individual's doctor decides on treatment, not the study sponsor (Astellas).

In this study, boys under 18 diagnosed with XLMTM will be followed for about 1 year. The health of their liver and gallbladder will be checked about every 6 weeks. This can be done at home, if preferred. A scan called a Fibroscan (also known as transient elastography) will check for signs of scarring in the liver (fibrosis) and the build-up of lipids. It is suggested that each boy will have a Fibroscan when they start the study and another scan when they complete the study.

This study will help understand liver, gallbladder, and bile duct issues in individuals with XLMTM over time. The goal is to improve their care and provide information to use in future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of XLMTM resulting from a genetically confirmed mutation in the MTM1 gene based on genetic test reports.
* Participant requires some mechanical ventilatory support (e.g., ranging from 24 hours per day full-time mechanical ventilation, to non-invasive support such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) during sleeping hours)
* Participant (as applicable) and/or parent(s)/carer is willing to comply with the recommended schedule of assessments.

Exclusion Criteria:

* Participant is currently enrolled in an interventional study designed to treat XLMTM.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 50 male participants < 18 years of age with genetically confirmed XLMTM will be enrolled at specialist sites.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of cholestasis | Up to Week 48
  Calculated as the number of new cases of cholestasis over 48 weeks divided by total duration of follow-up for enrolled participants.
Point prevalence of cholestasis | Day 1
  Point prevalence of cholestasis is defined as the proportion of participants who have had at least 1 case of cholestasis prior to Day 1 (baseline).
Prevalence of cholestasis | Up to 1 year
  Prevalence of cholestasis is defined as the proportion of participants who have had at least 1 case of cholestasis within 1 year of Day 1 (baseline).

SECONDARY OUTCOMES:
Genetic variants of MTM1 | Up to Week 48
  The association between genetic variants of MTM1 and cholestasis will be evaluated.
Risk of cholestasis temporarily associated with environmental modifiers | Up to Week 48
  Medication use, immunization history, infectious disease history and dietary habits will be collected.
Hospitalizations | Up to Week 48
  Frequency and reason for hospitalizations will be collected.
Duration of Hospitalizations | Up to Week 48
  Duration of hospitalization visits will be collected.
Emergency room visits | Up to Week 48
  Frequency and reason for visit will be collected.
Hepatology specialist visits | Up to Week 48
  Frequency and reason for visit will be collected.
Scheduled/unscheduled office visits | Up to Week 48
  Frequency and reason for visit will be collected.
Non-study-specified home healthcare visits | Up to Week 48
  Frequency and reason for visit will be collected.
Surgeries/procedures | Up to Week 48
  Frequency and type will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Gene Therapies
Locations (5):
- United States (5):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.